CLINICAL TRIAL: NCT06089590
Title: Ibd CAncer and seRious Infections in France (I-CARE 2)
Acronym: I-CARE 2
Status: Recruiting | Type: Observational
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Collaborators: Sanoia (Other)
Responsible Party: Sponsor
Other Study IDs: GETAID-2022-02
Record Dates: First submitted 2023-09-11; First posted 2023-10-18 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: IBD; Ulcerative Colitis; Crohn Disease
Keywords: UC; CD
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Group Anti-IL23p19: Patients treated with anti-IL23p19 (risankizumab, guselkumab, mirikizumab, brazikumab)
  Interventions: Other: Non-interventional
- Group Jak inhibitors: Patient treated with Jak inhibitors (tofacitinib, upadacitinib, filgotinib)
  Interventions: Other: Non-interventional
- Group S1P Modulators: Patient treated with S1P modulators (ozanimod, etrasimod)
  Interventions: Other: Non-interventional
- Group Anti TNF: Patient treated with anti-TNF (infliximab, adalimumab, golimumab) (with a maximal proportion of 25% as 1st first line biologic after conventional treatment (aminosalicylates, corticosteroids, thiopurines, methotrexate))
  Interventions: Other: Non-interventional
- Group Anti integrins: Patient treated with anti-integrins (vedolizumab)
  Interventions: Other: Non-interventional
- Group Anti IL12/23: Patient treated with anti-IL12/23 (ustekinumab)
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — This study is non-interventional, patients will be enrolled when initiating a treatment through standard of care procedures.

SUMMARY:
This is a French prospective longitudinal observational multicentre cohort study.

Primary objective : to assess prospectively the presence and the extent of safety concerns (cancer, serious infections, arterial and venous thrombotic events) in patients with CD and UC and treated with JAKi, anti-IL23p19, and S1p modulators.

DETAILED DESCRIPTION:
Number of patients : 6 000 at least Participating investigators : 250 at least

Recruitment period : 3 years 6 months

Primary objective : to assess prospectively the presence and the extent of safety concerns (cancer, serious infections, arterial and venous thrombotic events) in patients with CD and UC and treated with JAKi, anti-IL23p19, and S1p modulators.

Secondary objectives :

* To assess the presence and the extent of safety concerns in patients treated with JAKi, anti-IL23p19, and S1p modulators for each outcome of interest separately (cancer, serious infections, arterial thrombotic events, venous thrombotic events)
* To investigate prospectively the impact of JAKi, anti-IL23p19 and S1p modulators strategies on the natural history of IBD and their potential for disease modification by collecting validated surrogate markers such as mucosal healing and disease complications such as bowel damage (strictures, fistulas, abscess), surgeries, and hospitalizations
* To assess the evolution of ePROs on a trimester basis and the impact of JAKi, anti-IL23p19, and S1p modulators on ePROs in IBD
* To evaluate the benefit-risk ratio of strategies based on a wider use of JAKi, anti-IL23p19, and S1p modulators therapy for IBD
* To assess the healthcare costs and cost-efficacy of current therapeutic strategies in IBD.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an established diagnosis of Crohn's disease, ulcerative colitis or IBD unclassified based on usual radiological, endoscopic or histological criteria.
* Patient aged 18 and older accepting to sign the informed participating consent form, stating that he accepts to provide personal details (mobile and home phone number, e-mail address), to complete the e-PRO as required and to be contacted by a Study Coordinator and his gastroenterologist for the purpose of the study during the entire study period and during follow up if required.

Exclusion Criteria:

* Patient unable to sign the informed consent form
* Patient with no regular access to internet
* Patient refusing to sign the informed consent form
* Patient enrolled in a Randomized Clinical Trial (If the investigational product received was blinded, and if the treatment is unknown at time of enrolment in I-CARE 2)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBD patients initiating a biologic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2031-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of SAE declared by patients (cancer, serious infections, arterial and venous thrombotic events) | 4 to 7.5 years
  The primary objective of I-CARE 2 is to assess prospectively the presence and the extent of safety concerns (cancer, serious infections, arterial and venous thrombotic events) in patients with CD and UC and treated with JAKi, anti-IL23p19, and S1p modulators.
  The risk of cancers, serious infections and vascular events will be stratified according to IBD phenotype, disease activity (clinical, radiologic and endoscopic) and main comorbidities at baseline.

SECONDARY OUTCOMES:
Number of SAE declared by patients (cancer, serious infections, arterial and venous thrombotic events) | 4 to 7.5 years
  To assess the presence and the extent of safety concerns in patients treated with JAKi, anti-IL23p19, and S1p modulators for each outcome of interest separately
  * Cancer
  * Serious infections
  * Arterial thrombotic events
  * Venous thrombotic events
Treatment impact on IBD natural history | 4 to 7.5 years
  To investigate prospectively the impact of JAKi, anti-IL23p19 and S1p modulators strategies on the natural history of IBD and their potential for disease modification by collecting validated surrogate markers such as mucosal healing and disease complications such as bowel damage (strictures, fistulas, abscess), surgeries, and hospitalizations
ePRO | 4 to 7.5 years
  To assess the evolution of ePROs on a trimester basis and the impact of JAKi, anti-IL23p19, and S1p modulators on ePROs in IBD
Benefit-risk ratio | 4 to 7.5 years
  To evaluate the benefit-risk ratio of strategies based on a wider use of JAKi, anti-IL23p19, and S1p modulators therapy for IBD
Number and duration of hospitalization, surgery, endoscopy and other imaging | 4 to 7.5 years
  To assess the healthcare costs and cost-efficacy of current therapeutic strategies in IBD.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Kirchgesner, Principal Investigator — Hôpital Saint Antoine - APHP; Mathurin Fumery, Principal Investigator — CHU Amiens-Picardie
Locations (2):
- France (2):
  - CHU Amiens Picardie, Amiens
  - APHP Hôpital Saint Antoine, Paris

IPD SHARING:
Plan to Share IPD: No